CLINICAL TRIAL: NCT06262399
Title: Long-Term Follow-Up of Subjects Treated With NTLA 2002
Brief Title: Long-Term Follow-Up (LTFU) of Subjects Treated With NTLA 2002
Status: Enrolling by invitation | Type: Observational
Sponsor: Intellia Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: ITL-2002-CL-999; 2022-003778-22 (EudraCT Number)
Record Dates: First submitted 2024-01-12; First posted 2024-02-16 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-04

CONDITIONS: Hereditary Angioedema
MeSH Terms: conditions — Angioedemas, Hereditary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a follow-up study of subjects who received NTLA-2002 in a previous clinical trial as an observational evaluation of the long-term effects of the investigational therapy.

ELIGIBILITY:
Inclusion Criteria:

1. A subject has completed or discontinued from an Intellia-sponsored or -supported treatment protocol in which a complete or partial dose of NTLA-2002 was received.
2. A subject has provided informed consent for the LTFU study.
3. A subject is willing to attend study visits, complete protocol-required follow-up schedule, and comply with the study requirements.

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participating sites in an Intellia-sponsored clinical study of NTLA-2002.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2040-04 (Estimated); Study Completion 2040-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related Adverse Events (AEs); incidence of treatment-related Serious Adverse Events (SAEs); incidence of treatment-related Adverse Events of Special Interest (AESIs) defined per protocol | up to 15 years

SECONDARY OUTCOMES:
To evaluate the long-term efficacy of NTLA-2002 in previously treated subjects | up to 15 years
  Rate of Hereditary Angioedema (HAE) attacks overall and rate of HAE attacks requiring acute therapy. Total plasma kallikrein protein level.
Change from baseline in consumption of on-demand HAE medications for reported HAE attacks | up to 15 years
Change from baseline in healthcare utilization for HAE attacks | up to 15 years
Change from baseline in QoL parameters as measured by the MOXIE Angioedema-QoL instrument. | up to 5 years
Change from baseline in QoL parameters as measured by the EQ-5D-5L instrument. | up to 5 years
Change from baseline in QoL parameters as measured by the WPAI:GH instrument. | up to 5 years

CONTACTS AND LOCATIONS:
Locations (7):
- Campbelltown Hospital, Campbelltown, New South Wales, Australia
- France (2):
  - Centre National de Reference - Grenoble, Grenoble
  - Hôpital Claude Huriez, Lille
- Charite-Universitätsmedizin Berlin, Berlin, Germany
- University of Amsterdam Academic Medical Center, Amsterdam, Netherlands
- New Zealand Clinical Research, Auckland, New Zealand
- Cambridge University Hospitals NHS Foundation Trust, Addenbrooke's Hospital, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No